CLINICAL TRIAL: NCT04018976
Title: AVACEN Treatment Method and Postprandial Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Jeff Moore, Investigator, San Diego State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AVACENOGTT
Record Dates: First submitted 2019-07-06; First posted 2019-07-15 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Postprandial Hyperglycemia
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Heat and Vacuum (Experimental): AVACEN 100 applies heat and vacuum to hand
  Interventions: Device: AVACEN 100
- Heat Only (Active Comparator): AVACEN 100 applies heat only
  Interventions: Device: AVACEN 100 heat only
- Sham (Sham Comparator): AVACEN 100 applies neither heat nor vacuum
  Interventions: Device: AVACEN 100 sham

INTERVENTIONS:
Device: AVACEN 100 — The AVACEN 100 pulls a -30mmHg vacuum around the hand from the wrist down and applies heat (108 Fahrenheit) to the palm
  Arms: Heat and Vacuum
Device: AVACEN 100 heat only — The AVACEN 100 applies heat (108 Fahrenheit) to the palm
  Arms: Heat Only
Device: AVACEN 100 sham — The AVACEN 100 does not provide heat or vacuum
  Arms: Sham

SUMMARY:
A double-blind crossover randomized controlled trial to investigate the effects of the AVACEN device on postprandial blood glucose. The AVACEN device creates negative pressure around the hand while heating the palm. Two sham devices, one providing heat but no vacuum and one providing neither heat nor vacuum were also used. Each subject will use each of these three devices during the first hour of a 2-hour oral glucose tolerance test on separate visits. Subjects arrived in the morning following an overnight fast. Fasting blood glucose, blood pressure, tympanic temperature, and subjective thermal ratings were measured before and throughout the 2-hour oral glucose tolerance test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Diagnosis of diabetes, diabetes medication, hypertension medication

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Postprandial Blood Glucose | 30 minutes
  Measuring peak postprandial blood glucose with Contour Next glucometer

SECONDARY OUTCOMES:
Blood Pressure | 30 minutes
  Measuring blood pressure with automated cuff
Tympanic Temperature | 30 minutes
  Measuring tympanic temperature with infrared thermometer
ASHRAE 7 point thermal sensation scale | 30 minutes
  Measuring subjective temperature with thermal sensation scale

CONTACTS AND LOCATIONS:
Overall Officials: Jeff M Moore, B.S./B.S., Principal Investigator — San Diego State University
Locations (1):
- Jeff Moore, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No